CLINICAL TRIAL: NCT05780268
Title: A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients With COVID-19 (Trial H1: LY3819253 (LY-CoV555))
Brief Title: LY3819253 (LY-CoV555) for Inpatients With COVID-19 (An ACTIV-3/TICO Treatment Trial)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Network for Strategic Initiatives in Global HIV Trials (INSIGHT) (Network); University of Copenhagen (Other); Medical Research Council (Other Government); Kirby Institute (Other Government); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network); National Heart, Lung, and Blood Institute (NHLBI) (NIH); US Department of Veterans Affairs (U.S. Federal Agency); Prevention and Early Treatment of Acute Lung Injury (Other); Cardiothoracic Surgical Trials Network (Other); Eli Lilly and Company (Industry); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 014/ACTIV-3/H1
Record Dates: First submitted 2023-03-20; First posted 2023-03-22 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
Keywords: COVID-19; COVID 19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; SARS-CoV-2; SARS Coronavirus; ACTIV-3; ACTIV3; TICO
MeSH Terms: conditions — COVID-19; Coronaviridae Infections; Coronavirus Infections; RNA Virus Infections; Virus Diseases; Nidovirales Infections; Severe Acute Respiratory Syndrome | interventions — bamlanivimab; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3819253 plus SOC (Experimental): * LY3819253 7000 mg solution (10 vials of 20 mL solution containing 700 mg each); administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Biological: LY3819253; Biological: Remdesivir
- Placebo plus SOC (Placebo Comparator): * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Interventions: Biological: Placebo; Biological: Remdesivir

INTERVENTIONS:
Biological: LY3819253 — LY3819253 is a neutralizing immunoglobulin G (IgG)-1 monoclonal antibody (mAb) to the receptor binding domain (RBD) of the S protein of SARS-CoV-2
  Arms: LY3819253 plus SOC
Biological: Placebo — Commercially available 0.9% sodium chloride solution
  Arms: Placebo plus SOC
Biological: Remdesivir — Antiviral agent
  Other Names: Veklury

SUMMARY:
This study looks at the safety and effectiveness of LY3819253 in treating COVID-19 in people who have been hospitalized with the infection. Participants in the study will be treated with either LY3819253 plus current standard of care (SOC), or with placebo plus current SOC. This is ACTIV-3/TICO Treatment Trial H1.

DETAILED DESCRIPTION:
This is a treatment trial of the ACTIV-3/TICO master protocol (NCT04501978) to evaluate the safety and efficacy of LY3819253 in hospitalized patients infected with COVID-19.

This is a randomized, blinded, controlled sub-study of LY3819253 plus current standard of care (SOC) against placebo plus current SOC. The placebo arm may be shared across other sub-studies of the ACTIV-3/TICO master protocol. When more than one drug is being tested at the same time, participants will be randomly allocated to treatments or placebo.

Randomization will be stratified by study site pharmacy and disease severity. There are 2 disease severity strata: Participants without organ failure (severity stratum 1) and participants with organ failure (severity stratum 2).

An independent Data and Safety Monitoring Board (DSMB) will regularly review interim analyses and summarize safety and efficacy outcomes. The pace of enrollment with be initially restricted, and there will be an early review of safety data by the DSMB. At the outset of the trial, only participants in disease severity stratum 1 will be enrolled. This will continue until approximately 300 participants are enrolled and followed for 5 days. The exact number will vary according to the speed of enrollment and the timing of DSMB meetings. Prior to expanding enrollment to also include patients in disease severity stratum 2, safety will be evaluated and a pre-specified futility assessment by the DSMB will be carried out using 2 ordinal outcomes assessed at Day 5.

If LY3819253 passes the futility assessment, enrollment of participants will be expanded, seamlessly and without any data unblinding, to include participants in disease severity stratum 2 as well as those in disease severity stratum 1. Future interim analyses will be based on the primary endpoint of sustained recovery and will use pre-specified guidelines to determine early evidence of benefit, harm, or futility for the investigational agent. Participants will be followed for 18 months following randomization.

This trial will be conducted in several hundred clinical sites. Participating sites are affiliated with networks funded by the United States National Institutes of Health (NIH) and the US Department of Veterans Affairs.

ELIGIBILITY:
Inclusion Criteria: Refer to the master protocol (NCT04501978)

Exclusion Criteria: Refer to the master protocol (NCT04501978)

Additional Criteria:

Non-pregnant female participants who are of reproductive potential and male participants who are able to father a child must abstain from male/female sexual intercourse or agree to use two forms of effective contraception, where at least one form is highly effective (less than 1% failure rate), for the entirety of the study and for 90 days after investigational agent is administered. Highly effective methods of contraception (less than 1% failure rate) include, but are not limited to:

* combination oral contraceptives
* implanted contraceptives
* intrauterine devices

Effective methods of contraception include, but are not limited to:

* diaphragms and cervical caps with spermicide
* cervical sponges
* condoms with spermicide

NOTE:

* Use of male and female condoms as a double barrier method is not considered acceptable due to the high failure rate when these barrier methods are combined.
* Barrier protection methods without concomitant use of a spermicide are not an effective or acceptable method of contraception.
* Periodic abstinence (e.g., calendar, ovulation, symptothermal, postovulation methods), and withdrawal are not acceptable methods of contraception. Participants not of reproductive potential are eligible without requiring the use of a contraceptive method. Participant-reported history is acceptable documentation of surgical sterilization and menopause. Participants with pregnant partners should use condoms during vaginal intercourse through 90 days after investigational agent administration. Participants should refrain from sperm donation through 90 days after investigational agent administration. NOTE: Reproductive potential is defined as patients who have reached menarche, who have not been post-menopausal for at least 12 consecutive months with follicle-stimulating hormone (FSH) ≥ 40 IU/ml or 24 consecutive months if an FSH is not available, who have not undergone surgical sterilization, who do not have other clinical condition that could induce amenorrhea, who are not taking medications such as oral contraceptives, hormones, gonadotropin releasing hormone, antiestrogens, selective estrogen receptor modulators (SERMs) or chemotherapy that could induce amenorrhea. Individuals with permanent infertility due to an alternate medical cause (e.g. Mullerian agenesis, androgen insensitivity), investigator discretion should be applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Lundgren, Prof., Principal Investigator — INSIGHT Copenhagen International Coordinating Centre, Rigshospitalet, University of Copenhagen; James Neaton, Prof., Study Chair — INSIGHT Statistical and Data Management Center, University of Minnesota
Locations (57):
- United States (42):
  - Banner University Medical Center Tucson (Site 206-004), 1625 N. Campbell Avenue, Tucson, Arizona
  - Community Regional Medical Center (Site 203-005), 2823 Fresno Street, Fresno, California
  - Keck Hospital of USC (Site 301-020), 1500 San Pablo Street, Los Angeles, California
  - UCSF Medical Center at Mount Zion (Site 203-007), 1600 Divisadero St., San Francisco, California
  - San Francisco VAMC (Site 074-002), 4150 Clement St., San Francisco, California
  - UCSF Medical Center (Site 203-001), Moffitt-Long Hospital, 505 Parnassus Ave., San Francisco, California
  - Stanford University Hospital & Clinics (Site 203-003), 300 Pasteur Dr., Stanford, California
  - University of Colorado Hospital (Site 204-001), 12605 E. 16th Avenue, Aurora, Colorado
  - Denver Public Health (Site 017-004), 660 Bannock St., MC2600 (Infectious Disease Clinic), Denver, Colorado
  - MedStar Georgetown University Hospital (Site 067-001), 3800 Reservoir Road NW, Washington D.C., District of Columbia
  - Miami VAMC (Site 074-003), 1201 NW 16 Street, Miami, Florida
  - Emory University (Site 301-008), The Emory Clinic, Bldg. A, Suite 2236, 1365 Clifton Rd., NE, Atlanta, Georgia
  - University of Kentucky Hospital (Site 210-004), 1000 South Limestone St., Lexington, Kentucky
  - Ochsner Clinic Foundation (Site 301-015), 1514 Jefferson Highway, New Orleans, Louisiana
  - University of Maryland Medical Center (Site 301-019), 22 South Greene Street, Baltimore, Maryland
  - Massachusetts General Hospital (Site 202-002), 55 Fruit Street, Boston, Massachusetts
  - Baystate Medical Center (Site 201-001), 759 Chestnut Street, Springfield, Massachusetts
  - University of Michigan (Site 205-001), 1500 East Medical Center Drive, Ann Arbor, Michigan
  - Henry Ford Health System, Henry Ford Hospital (Site 014-001), 2799 W. Grand Blvd., Detroit, Michigan
  - Hennepin Healthcare (Site 027-001), 701 Park Avenue, Minneapolis, Minnesota
  - University of Mississippi Medical Center (Site 202-005), 2500 North State Street, Jackson, Mississippi
  - Dartmouth-Hitchcock Medical Center/Mary Hitchcock Memorial Hospital (Site 301-024), One Medical Center Drive, Lebanon, New Hampshire
  - Montefiore Medical Center Weiler Hospital (Site 206-003), 1825 Eastchester Road, The Bronx, New York
  - Montefiore Medical Center Moses Hospital (Site 206-001), 111 E. 210th Street, The Bronx, New York
  - Duke University Hospital (Site 301-006), 2301 Erwin Road, Durham, North Carolina
  - Wake Forest University Health Sciences (Site 210-001), Medical Center Blvd, Winston-Salem, North Carolina
  - Cleveland Clinic Fairview Hospital (Site 207-005), 18101 Lorain Avenue, Cleveland, Ohio
  - Cleveland Clinic Foundation (Site 207-001), 9500 Euclid Avenue, Cleveland, Ohio
  - Cleveland Clinic Marymount Hospital (Site 207-006), 12300 McCraken Road, Garfield Heights, Ohio
  - Oregon Health & Science University (Site 208-003), 3181 SW Sam Jackson Park Rd., Portland, Oregon
  - Vanderbilt University Medical Center (Site 212-001), 1211 Medical Center Drive, Nashville, Tennessee
  - UT Southwestern Medical Center (Site 084-001), 1936 Amelia Court, 2nd Floor, Dallas, Texas
  - Baylor, Scott and White Health (Site 301-003), Baylor University Medical Center, 3500 Gaston Ave., Dallas, Texas
  - Memorial Hermann Hospital (Site 203-006), 6411 Fannin Street, Houston, Texas
  - Michael E. DeBakey Veterans Affairs Medical Center (MEDV AMC) (Site 074-006), 2002 Holcombe Blvd., Houston, Texas
  - Intermountain Medical Center (Site 211-001), 5121 South Cottonwood Street, Murray, Utah
  - University of Utah Hospital (Site 211-002), 419 Wakara Way, Suite 207, Salt Lake City, Utah
  - University of Virginia Health Systems (Site 301-021), 1215 Lee Street, Charlottesville, Virginia
  - Virginia Commonwealth University Health System (Site 210-005), 1250 East Marshall Street, Richmond, Virginia
  - Harborview Medical Center (Site 208-001), 325 9th Avenue, Seattle, Washington
  - University of Washington Medical Center - Montlake (Site 208-006), 1959 NE Pacific Street, Seattle, Washington
  - West Virginia University (Site 301-023), One Medical Center Drive, Morgantown, West Virginia
- Denmark (8):
  - Aalborg Hospital (Site 625-005), Hobrovej 18, Aalborg
  - Aarhus Universitetshospital, Skejby (Site 625-002), Department of Infectious Diseases, Palle Juul-Hensens Boulevard 99, Aarhus N
  - Righospitalet (Site 625-006), Blegdamsvej 9,, Copenhagen Ø
  - Herlev/Gentofte Hospital (Site 625-012), Medicinsk Afdeling, Herlev Ringvej 75, Herlev
  - Nordsjællands Hospital (Site 625-009), Dyrehavevej 29, Hillerød
  - Hvidovre University Hospital, Department of Infectious Diseases (Site 625-001), Kettegård allé 30, Hvidovre
  - Kolding Sygehus (Site 625-011), Medicinsk Afdeling, Sygehusvej 24, Kolding
  - Odense University Hospital (Site 625-004), Infektionsmedicinsk Forskningsenhed, J.B. Winsløwsgade 4, Odense
- Tan Tock Seng Hospital (Site 612-201), National Centre for Infectious Diseases (NCID), 11 Jalan Tan Tock Seng, Singapore, Singapore
- Spain (6):
  - Hospital Universitari Germans Trias i Pujol (Site 626-003), Infectious Disease Unit, Second Floor, Building Maternal, Road Canyet s/n, Badalona, Barcelona
  - Hospital Del Mar (Site 626-025), Paseo Maritimo 25-29, Barcelona
  - Hospital Clínic de Barcelona (Site 626-004), Carrer de Villaroel 170, Barcelona
  - Hospital General Universitario Gregorio Marañón (Site 626-001), Dr. Esquerdo, 46, Madrid
  - Hospital Clínico San Carlos (Site 626-017), Enfermedades infecciosas, C/Martin Lagos CN, Madrid
  - UCICEC (Clinical Trial Unit) Hospital Universitario La Paz (Site 626-012), Paseo de la Castellana 261, 2a planta Hospital Maternal, Madrid

REFERENCES:
- [Result] ACTIV-3/TICO LY-CoV555 Study Group; Lundgren JD, Grund B, Barkauskas CE, Holland TL, Gottlieb RL, Sandkovsky U, Brown SM, Knowlton KU, Self WH, Files DC, Jain MK, Benfield T, Bowdish ME, Leshnower BG, Baker JV, Jensen JU, Gardner EM, Ginde AA, Harris ES, Johansen IS, Markowitz N, Matthay MA, Ostergaard L, Chang CC, Davey VJ, Goodman A, Higgs ES, Murray DD, Murray TA, Paredes R, Parmar MKB, Phillips AN, Reilly C, Sharma S, Dewar RL, Teitelbaum M, Wentworth D, Cao H, Klekotka P, Babiker AG, Gelijns AC, Kan VL, Polizzotto MN, Thompson BT, Lane HC, Neaton JD. A Neutralizing Monoclonal Antibody for Hospitalized Patients with Covid-19. N Engl J Med. 2021 Mar 11;384(10):905-914. doi: 10.1056/NEJMoa2033130. Epub 2020 Dec 22. PMID 33356051

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from 31 sites in 3 countries (Denmark, Singapore, USA). The first subject was enrolled on 5 Aug 2020 and the last subject was enrolled on 13 Oct 2020.
Groups:
- LY3819253 Plus SOC: * LY3819253 7000 mg solution (10 vials of 20 mL solution containing 700 mg each); administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  LY3819253: LY3819253 is a neutralizing immunoglobulin G (IgG)-1 monoclonal antibody (mAb) to the receptor binding domain (RBD) of the S protein of SARS-CoV-2
  Remdesivir: Antiviral agent
- Placebo Plus SOC: * Placebo administered by IV infusion
  * Remdesivir is provided to all study participants as SOC unless contraindicated for an individual patient; administered by IV infusion
  Placebo: Commercially available 0.9% sodium chloride solution
  Remdesivir: Antiviral agent
Period: Overall Study
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Started | 163 | 151
Completed | 163 | 151
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC | Total
Number analyzed (Participants) | 163 | 151 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (14.2) | 58.9 (16.3) | 59.6 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 71 | 137
  Male | 97 | 80 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 33 | 74
  Not Hispanic or Latino | 122 | 118 | 240
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 3 | 0 | 3
  Race: Asian | 6 | 7 | 13
  Race: Native Hawaiian or Pacific Islander | 1 | 1 | 2
  Race: Black or African American | 32 | 34 | 66
  Race: White | 90 | 88 | 178
  Race: More than one race | 1 | 1 | 2
  Race: Other | 4 | 4 | 8
  Race: Only ethnicity reported | 26 | 16 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Sustained Recovery
Description: Sustained recovery defined as being discharged from the index hospitalization, followed by being alive and home for 14 consecutive days prior to Day 90.
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants | 144 | 136

2. Primary Outcome: Number of Participants With an Ordinal Outcome on Day 5
Description: Ordinal outcome with 7 mutually exclusive categories
Time Frame: Status on Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants
  7 = Death | 1 | 0
  6 = Invasive ventilation, ECMO, mechanical circulatory support, new renal replacement therapy | 8 | 5
  5 = Non-invasive ventilation or high flow oxygen | 24 | 22
  4 = Supplement oxgen (≥4 L/min or ≥4 L/min above baseline, but not high flow oxygen) | 18 | 11
  3 = Supplement oxgen (<4 L/min or <4 L/min above baseline, but not high flow oxygen) | 30 | 33
  2 = Limiting symptoms due to COVID-19, but not need of new or increased oxygen from baseline | 51 | 45
  1 = No limiting symptoms due to COVID-19 | 31 | 35

3. Secondary Outcome: Number of Participants Who Died From All Causes
Description: All-cause mortality
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants | 13 | 11

4. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 5
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 5
Time Frame: Through Day 5
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants | 45 | 28

5. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 28
Description: Death, SAE, clinical organ failure, serious infections, or Grade 3 or 4 event through Day 28
Time Frame: Through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants | 52 | 42

6. Secondary Outcome: Number of Participants With a Safety Outcome Through Day 90
Description: Death, SAE, clinical organ failure, serious infections through Day 90
Time Frame: Through Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
Number analyzed (Participants) | 163 | 151
Participants | 45 | 41

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | LY3819253 Plus SOC | Placebo Plus SOC
All-Cause Mortality (participants affected / at risk) | 13/163 | 11/151
Serious Adverse Events (participants affected / at risk) | 9/163 | 12/151
Other Adverse Events (participants affected / at risk) | 41/163 | 27/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3819253 Plus SOC (N=163) | Placebo Plus SOC (N=151)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponataemis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic obstructive pulonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypotension (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY3819253 Plus SOC (N=163) | Placebo Plus SOC (N=151)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pancreatitits (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 9 (10) | 5 (5)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Odema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 2 (3) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Pseudomonas infection (Infections and infestations) | 1 (1) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
10016803 (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoglyceamia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Dizzyness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0)
Panic attack (Nervous system disorders) | 1 (1) | 0 (0)
Mental status changes (Nervous system disorders) | 7 (7) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 5 (7) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 10 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pneumoththorax (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 6 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Trial H1 Protocol (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT05780268/Prot_000.pdf
  • Study Protocol: Master Protocol (2021-08-17): https://cdn.clinicaltrials.gov/large-docs/68/NCT05780268/Prot_003.pdf
  • Statistical Analysis Plan (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT05780268/SAP_001.pdf
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT05780268/ICF_002.pdf